CLINICAL TRIAL: NCT01709552
Title: A Computer-based Intervention for Women With Substance Use and Intimate Partner Violence in the Emergency Department
Brief Title: Brief Intervention for Substance Use and Partner Abuse Among Females in the ER
Acronym: B-SAFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Esther Choo, Assistant Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K23DA031881-02 (NIH)
Record Dates: First submitted 2012-08-10; First posted 2012-10-18 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Substance Related Disorders; Domestic Violence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer Intervention (Experimental): Patients randomized to the computer intervention will complete the B-SAFER computer program during their emergency department visit.
  Interventions: Behavioral: Computer Intervention
- Control (Sham Comparator): Patients randomized to the control arm will receive a time-equivalent computer-based program unrelated to substance use or partner violence.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Computer Intervention — Patients randomized to the computer intervention will complete the B-SAFER computer program during their emergency department visit.
  Arms: Computer Intervention
Behavioral: Control — Patients randomized to the control arm will receive a time-equivalent computer-based program unrelated to substance use or partner violence.
  Arms: Control

SUMMARY:
The purpose of this study is to target co-occurring problems of substance use and intimate partner violence (IPV) using a computer-based intervention, B-SAFER (Brief intervention for Substance use and partner Abuse for Females in the Emergency Room). This project will develop and test the computer-based intervention, examining primary outcomes of substance use and utilization of relationship safety resources.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* English or Spanish language proficiency sufficient to understand and complete study procedures
* moderate drug use in the prior 3 months (by NM-ASSIST)
* IPV victimization in the prior 6 months (by WAST)
* access to a phone

Exclusion Criteria:

Patients who are:

* intoxicated
* medically unstable as determined by ED staff
* suicidal ideation
* psychosis
* combative
* in police custody

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in past-month drug use days | 1 month, 3 month
  Drug use based on Timeline Followback.
Change in use of relationship safety behaviors and referral resources for IPV. | 2 weeks, 1 month, 3 months
  Based on Safety Behavior Checklist and Effectiveness in Obtaining Resources scales.

SECONDARY OUTCOMES:
Change in readiness to change drug use. | 2 week, 1 month, 3 months
  Based on readiness to change rulers.
Change in readiness to change scale for relationship safety behaviors. | 2 weeks, 1 month, 3 months
  Based on readiness to change rulers.

CONTACTS AND LOCATIONS:
Overall Officials: Esther K Choo, MD MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital Department of Emergency Medicine, Providence, Rhode Island, United States